CLINICAL TRIAL: NCT03322514
Title: Effect of Increased Colonic Propionate on Weight Loss During a Hypo-caloric Diet.
Brief Title: Colonic Propionate, Appetite, and Weight Loss
Acronym: ProAp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16HH3560; 210536 (Other: IRAS)
Record Dates: First submitted 2017-05-10; First posted 2017-10-26 (Actual); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Healthy Obesity, Metabolically; Appetite Regulation
Keywords: gut hormones; obesity; appetite; propionate; fermentation
MeSH Terms: conditions — Obesity, Metabolically Benign; Obesity | interventions — Inulin

STUDY DESIGN:
Intervention Model Description: double blind, randomised, controlled, paralleled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 10 g of Inulin-Propionate Esters will be administered per day
  Interventions: Dietary Supplement: Inulin-Propionate Esters
- Inulin (Active Comparator): 10 g of Inulin will be administered per day
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin-Propionate Esters — Inulin (β(2-1) linked polymer of fructose) carrier with an ester linked to propionate (propionate ester). Thus, propionate is only released when the carrier molecule inulin is fermented by colon microflora.
  Arms: experimental group
Dietary Supplement: Inulin — Inulin
  Arms: Inulin

SUMMARY:
The current protocol aims to investigate the impact of the propionate ester in conjugation with restricted diet on appetite and weight loss.

DETAILED DESCRIPTION:
DIET AND OBESITY:

Obesity has reached epidemic proportions worldwide. In the United Kingdom, 58% of adult women and 65% of adult men are either overweight or obese (Health and Social Care Information Centre 2014), with the expectation that rates will increase (Ng et al. 2014). Obesity, mainly caused by a chronic positive energy balance, is a known risk factor that contributes to the development of type 2 diabetes and cardiovascular diseases, and the subsequent morbidities and mortalities (Kopelman 2007). A positive energy balance is inevitable with the composition of current western diet that contain refined (fibre-depleted) carbohydrates that are consumed quickly, and have minimal effects on long-term satiety (Cleave 1974; Heaton 1973).

NONDIGESTIBLE CARBOHYDRATES:

The quality and quantity of diet has changed dramatically over the last fifty years. Of which, carbohydrates have the most significant changes; from unprocessed fruits and vegetables based carbohydrates to more processed cereal based ones (Cordain et al. 2005). Epidemiological studies have shown that, as a result, ancestral diets had greater amounts of Non-Digestible Carbohydrates (NDC) than modern diets (>100g/day compared to <15g/day) with the inclusion of more indigestible intact cell wall plant material, such as tubers, grasses and sedges (Eaton 2006). A strong association has been established between increased weight gain with decreased NDC intake (Liu et al. 2003). Furthermore, increasing intake of NDC have shown to induce satiety and improve body composition in animals (So et al. 2007) and humans (Bouché et al. 2002).

LOW CALORIC HIGH NDC DIET IN LOSING WEIGHT Applying energy-restricted diets is one of the first steps to treat obesity. However, weight regain in weight maintenance period could happen due to resting energy expenditure reduction and lean mass loss. The inclusion of specific foods to the nutritional intervention is being investigated in order to produce persistent weight losses (Abete et al. 2008). It was suggested earlier that the addition of high fibre NDC foods to a hypocaloric diet would help reducing the incidence of metabolic syndrome and increasing the dietary compliance (Hermana et al, 2011). The high fibre content in combination with a low glycemic index diet, can both result in higher satiety effects with an increased mitochondrial oxidation, all favour weight loss.

PROPIONATE AND THE FFAR2 RECEPTOR:

Production of short chain fatty acids (SCFA) is the main by-product of NDC colonic fermentation (Pawlak et al. 2004). Of them, colonic propionate was found to play a critical role directly in the colon and systematically after its absorption into the circulation (Wong et al. 2006). Free Fatty Acid Receptor 2 (previously known as orphan G-coupled Protein Receptor 43) has been discovered to has high affinity to propionate (Brown et al. 2003). It is expressed on the distal ileum and colon L-enteroendocrine cells (Karaki et al. 2008), adipocytes and certain monocytes lineage (Hong et al. 2005).

THE ROLE OF PROPIONATE IN GUT HORMONE RELEASE AND APPETITE REGULATION:

The L-enteroendocrine colonic cells are responsible of secreting anorexic gut hormones (PYY and GLP-1) physiologically in response to food. These hormones are capable of inducing satiety through signalling the brain appetite centre (Murphy & Bloom 2006). Propionate-induced FFAR2 activation have found to cause the release of these hormones in vitro. Moreover, NDC ingestion was found to stimulate the release of these hormones in animals, resulting in decreasing food ingestion (Delzenne et al. 2005). Propionate was shown to replicate the same effects in further studies, suggesting the owning of the beneficial effects of NDC on appetite and gut hormones to propionate production.

SHORT CHAIN FATTY ACID ESTER:

Administering NDCs that promote the production of propionate is an attractive way to increase the level of propionate over an extended period of time. However, due to variability of the gut microbita activity, administering high proportions (≥ 35g/d) of dietary fibres in human diets to increase colonic propionate does not reliably or predictably provide the same SCFA levels in colon or systemically (Cummings 1981). Oral propionate supplementation is another method, but unfortunately its short plasma half-life, poor palatability, and the fact that its main absorption happens in the small intestine limit its use as a food supplement (Frost et al. 2003).

A novel system has been developed by Dr Douglas Morrison, (Scottish Universities Environmental Research Centre (SUERC)). This molecule of inulin (β(2-1) linked polymer of fructose) carrier with an ester linked to propionate (propionate ester) was demonstrated to reliably and reproducibly increase colonic propionate while prevent the side effects of NDC (Chambers et al. 2015). Thus, propionate is only released when the carrier molecule inulin is fermented by colon microflora, which was estimated to be 180 minutes post-ingestion. (Chambers et al. 2014). Chambers et al. (2015) were able to show that 10g of Inulin-Propionate Esters (IPE) has the ability to deliver 2.4g of propionate to the colon, that is an increment of 2.5-fold of propionate production in the colon, a level that is achieved only with 60g/d via traditional dietary fibre supplementation. The same group has also demonstrated that while the acute administration of this supplement caused increments in Plasma GLP-1 and PYY and reduced food ingestion, the long term (24 weeks) supplementation of propionate ester significantly reduced body weight gain and the development of abdominal adipose tissue (Chambers et al. 2014). Interestingly, none of the long term participants reported any side effects from the intake of propionate esters. Increasing colonic propionate is, therefore, one of the attractive strategies to manage weight and diabetes risk factors.

The current protocol aims to investigate the impact of the propionate ester in conjugation with restricted diet on appetite and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese ((BMI) of 25-35 kg/m2)
* healthy
* aged between 18 and 65 years

Exclusion Criteria:

* Weight change of ≥ 3kg in the preceding 2 months
* Undergone any weight loss surgery or gastric procedures to promote weight loss
* Current smokers
* Substance abuse
* Excess alcohol intake
* Pregnancy
* Diabetes
* Cardiovascular disease
* Cancer
* Gastrointestinal disease e.g. inflammatory bowel disease or irritable bowel syndrome
* Kidney disease
* Liver disease
* Pancreatitis
* Use of medications likely to interfere with energy metabolism, appetite regulation and hormonal balance, including: anti-inflammatory drugs or steroids, antibiotics, androgens, phenytoin, erythromycin or thyroid hormones.

Any participants with the above conditions would already have an altered pattern of hormones and inflammatory molecules because of their disease process and would therefore give us confounding or misleading results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Frost, Principal Investigator — Dietitian; PhD in Nutrition; Professor of nutrition and dietetics
Locations (1):
- NIHR/Wellcome Trust Imperial Clinicial Research Facility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] M. Khatib, E. Chambers, D. Morrison and G. Frost. A pilot study to evaluate the effect of increased colonic propionate on appetite during a hypocaloric diet. Proceedings of the Nutrition Society (2018), 77 (OCE4), E119.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Group | Inulin
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Inulin | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (5.9) | 35.2 (12.1) | 33.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight Loss Compared to Baseline
Description: The weight assessed by a body scale
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: kg
Groups:
- Experimental Group: 10 g of Inulin-Propionate Esters administered per day
- Inulin: 10 g of Inulin administered per day
Arm/Group | Experimental Group | Inulin
Number analyzed (Participants) | 5 | 5
kg | -2.6 (0.9) | -3 (1.04)
Statistical Analysis 1: Comparison: Experimental Group vs Inulin; Test type: Superiority; p = 0.8, t-test, 2 sided
Statistical Analysis 2: Comparison: Experimental Group; Baseline to 12 weeks; Test type: Superiority; p = 0.04, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin; Baseline to 12 weeks; Test type: Superiority; p = 0.1, t-test, 2 sided

2. Secondary Outcome: Glucose Blood Level Baseline to 12 Weeks
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Experimental Group | Inulin
Number analyzed (Participants) | 5 | 5
mmol/L
  Baseline | 4.9 (0.1) | 4.4 (0.1)
  12 weeks | 5.1 (0.1) | 4.8 (0.1)
Statistical Analysis 1: Comparison: Experimental Group vs Inulin; Test type: Superiority; p = 0.8, ANOVA
Statistical Analysis 2: Comparison: Experimental Group; Baseline to 12 weeks; Test type: Superiority; p = 0.3, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin; Baseline to 12 weeks; Test type: Superiority; p = 0.3, t-test, 2 sided

3. Secondary Outcome: Insulin Level in Serum
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Error); unit: mU/mL
Arm/Group | Experimental Group | Inulin
Number analyzed (Participants) | 5 | 5
mU/mL
  Baseline | 50.4 (10.8) | 48.9 (18.3)
  12 weeks | 41.0 (6.7) | 46.0 (21.1)
Statistical Analysis 1: Comparison: Experimental Group vs Inulin; Test type: Superiority; p = 0.9, ANOVA
Statistical Analysis 2: Comparison: Experimental Group; Baseline to 12 weeks; Test type: Superiority; p = 0.4, t-test, 2 sided
Statistical Analysis 3: Comparison: Inulin; baseline to 12 weeks; Test type: Superiority; p = 0.7, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Experimental Group | Inulin
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT03322514/Prot_SAP_000.pdf